CLINICAL TRIAL: NCT05198362
Title: A Phase 2b, Double-blind, Randomized, Placebo-controlled, Multi-center, 16-week Dose Finding, Safety and Efficacy Study With Open-label Extension (OLE) Period of Tesomet in Subjects With Prader-Willi Syndrome
Brief Title: Study of Tesomet With Open-label Extension in Subjects With Prader-Willi Syndrome
Acronym: PWS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to financial considerations Sponsor is unable to complete the trial and assess the planned objectives/endpoints. No subjects have been randomized to treatment in the clinical trial and the decision therefore has no safety concern for patients
Sponsor: Saniona (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TM006
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Prader-Willi Syndrome
Keywords: hyperphagia
MeSH Terms: conditions — Prader-Willi Syndrome; Hyperphagia | interventions — Tesofensine; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Once-daily PO for 16 weeks during the double-blind period; then if eligible for OLE, once-daily dosing for 36 weeks of the highest tolerated Tesomet dose from the double-blind period
  Interventions: Other: Placebo; Drug: Tesomet
- Tesomet Low Dose (Experimental): Once-daily PO for 16 weeks during the double-blind period; then if eligible for OLE, once-daily dosing for 36 weeks of the highest tolerated dose from the double-blind period
  Interventions: Drug: Tesomet
- Tesomet Medium Dose (Experimental): Once-daily PO for 16 weeks during the double-blind period; then if eligible for OLE, once-daily dosing for 36 weeks of the highest tolerated dose from the double-blind period
  Interventions: Drug: Tesomet
- Tesomet High Dose (Experimental): Once-daily PO for 16 weeks during the double-blind period; then if eligible for OLE, once-daily dosing for 36 weeks of the highest tolerated dose from the double-blind period
  Interventions: Drug: Tesomet

INTERVENTIONS:
Other: Placebo — Inactive comparator
  Arms: Placebo
Drug: Tesomet — Fixed-dose combination
  Other Names: tesofensine; metoprolol

SUMMARY:
This study will evaluate the safety and efficacy of Tesomet (tesofensine + metoprolol) in subjects with PWS.

DETAILED DESCRIPTION:
For the double-blind portion of the study, dosing will be initiated in a subgroup of adults who are 18-65 years of age. Following independent Data Monitoring Board review of subgroup safety data, and review and confirmation to proceed by FDA, enrollment of subjects <18 years of age will commence.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject and their legally authorized representative must be willing to provide informed consent
* Confirmed genetic diagnosis of PWS
* Body mass index (BMI) within the following range at Screening:

  1. Female and male subjects 18 to 65 years of age: 27 to 60 kg/m2; or
  2. Female and male subjects 13 to 17 years of age with BMI that is at least 85th percentile for age and sex;
* Female subjects must be of non-child-bearing potential
* Documented stable body weight
* Moderate hyperphagia at Screening and at Baseline
* Participants must have a reliable and stable caregiver who should be able to spend an adequate amount of time with the participants to be able to address behaviors, activities and symptoms
* Male subjects who are sexually active must be surgically sterile

Key Exclusion Criteria:

* Females who are pregnant, breastfeeding, or actively intending to become pregnant during the study
* Sitting BP that meets the following criteria after 5 minutes of rest at Screening:

  1. Adult subjects with systolic BP >/=145 mmHg or <100 mmHg; or
  2. Adult subjects with diastolic BP >/=95 mmHg or <70 mmHg; or
  3. Adolescent subjects with a systolic or diastolic BP that is 95th percentile or greater for age and sex
* Type 1 diabetes mellitus
* History of dementia (eg, Alzheimer's disease, Parkinson's disease)
* History of bulimia or anorexia nervosa
* History of major depressive disorder within 2 years prior to Screening, or any history of other severe psychiatric disorder (eg, schizophrenia, bipolar disorder), or symptoms of delusions, hallucinations, or mania/hypomania within 90 days prior to Screening, as described by the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5)
* Uncontrolled endocrine disorders (eg, Cushing syndrome, Addison's, hypothyroidism, hyperthyroidism)
* Medical condition or recent systemic infection that, in the opinion of the Investigator, could impact the safety of the subject
* Use of prohibited medications, including current use of SSRIs/SNRIs

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Hyperphagia | Baseline to Week 16
  Change in Hyperphagia Questionnaire for Clinical Trials (HQ-CT) total score

SECONDARY OUTCOMES:
Change in Body Weight | Baseline to Week 16
  Percentage change in body weight
Hyperphagia Severity (Caregiver) | Baseline to Week 16
  Change in caregiver rating of hyperphagia severity
Hyperphagia Change (Caregiver) | Week 16
  Proportion of caregiver responses for change in subject's hyperphagia
PWS Severity (Clinician) | Baseline to Week 16
  Change in clinician rating of the subject's PWS severity
Overall Status Change (Clinician) | Week 16
  Proportion of clinician responses for change in subject's overall clinical status

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Guillaume, MS, Study Director — Saniona
Locations (1):
- Sparrow Clinical Research Institute, Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The Sponsor will consider requests from qualified researchers for access to TM006 study materials
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following completion of Tesomet clinical development